CLINICAL TRIAL: NCT03464591
Title: Cardiac Speckle Tracking Myocardial Strain Balance Method: a New Method to Evaluate the Effect of Pulmonary Hypertension on the Prognosis
Brief Title: Cardiac Speckle Tracking Myocardial Strain Balance
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: echocardiography of PH
Record Dates: First submitted 2018-03-07; First posted 2018-03-14 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2017-11

CONDITIONS: Pulmonary Hypertension; Echocardiography
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators intend to evaluate the function of left heart and right heart and the motion balance between four chambers of the heart by speckle tracking technique during the follow-up of patients with pulmonary hypertension, and explore the relationship between the balance and prognosis of patients.

DETAILED DESCRIPTION:
Pulmonary hypertension is a fatal disease with progressive progressive vascular resistance that leads to the loss of right heart function. Right heart failure is the cause of death in most patients with end-stage pulmonary hypertension, and right heart function is also an important factor in determining the prognosis of patients.

Echocardiography speckle tracking technology is a noninvasive technique for evaluating global and local cardiac function by tracking myocardial ultrasonic spots through computer image analysis technology and quantifying myocardial deformation.

The investigators intend to evaluate the function of left heart and right heart and the motion balance between four chambers of the heart by speckle tracking technique during the follow-up of patients with pulmonary hypertension, and explore the relationship between the balance and prognosis of patients.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed with pulmonary hypertension by right cardiac catheterization The patient is between 18-80 years of age The date of diagnosis was from 2007 to 2017

Exclusion Criteria:

Cardiomyopathy Severe complications Pregnancy Atrial fibrillation, or other irregular heart rhythm Poor ultrasonic image quality

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From 2007 to date, 18-80 year old patients with mean pulmonary arterial pressure ≥25mmHg measured by right heart catheterization
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
outcome | one year
  death or time out

CONTACTS AND LOCATIONS:
Overall Officials: Shen Jieyan, PhD, Study Chair — RenJi Hospital, School of Medicine, Shanghai Jiaotong University; Shen Xuedong, PhD, Study Chair — RenJi Hospital, School of Medicine, Shanghai Jiaotong University
Locations (1):
- Renji Hospital, Shanghai, China